CLINICAL TRIAL: NCT05534113
Title: Sequential Envafolimab Immunotherapy After Patients With ctDNA EGFR Mutation Clearance by Treatment With Almonertinib in EGFR-Mutant, PD-LI Positive Non-small-cell Lung Cancer：Efficacy and Safety Clinical Trial
Brief Title: Envafolimab Immunotherapy After ctDNA EGFR Clearance by Treatment With Almonertinib in EGFR-Mutant, PD-LI Positive NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yongqian Shu, Study Principal Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-439
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EGFR; ctDNA; PD-L1; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sequential Envafolimab therapy after Almonertinib treatment (Experimental): Sequential Envafolimab therapy after patients with ctDNA EGFR mutation clearance and achieve stable radiographically deep response after treatment with Almonertinib
  Interventions: Drug: Almonertinib Envafolimab

INTERVENTIONS:
Drug: Almonertinib Envafolimab — Subjects will receive Almonertinib treatment for 6-8 weeks after enrollment, and receive ctDNA detection and radiography assessment again.
  If the EGFR mutation is positive, according to the patient's condition and clinical actual situation, subjects will receive combination therapy scheme, follow-up once every 6 weeks. The treatment will continue until the disease progress assessed by radiography.
  If the EGFR mutation turns negative and stable radiographically deep response, stop Almonertinib treatment and receive the relevant assessment before immunotherapy and receive Envafolimab treatment，and follow-up once every 6 weeks. The treatment of Envafolimab will continue until the EGFR mutation is positive again or disease progress assessed by radiography.

SUMMARY:
This is a prospective, single-arm, open-label, interventional clinical study, aimed at exploring the efficacy and safety of sequential Envafolimab immunotherapy after patients with ctDNA EGFR mutation clearance and achieved stable radiographically deep esponse after first line treatment with Almonertinib in EGFR-Mutant, PD-LI positive non-small-cell lung cancer.

DETAILED DESCRIPTION:
The study includes a screening period (not more than 28 days after the subject signs informed consent to before the first medication), treatment period (including Almonertinib treatment in 6-8 weeks after enrollment\ctDNA testing and radiographically imaging assessment\ctDNA guiding sequential Envafolimab immunotherapy) and follow-up period (including survival and safety) .

Eligible subjects receive 110 mg of Almonertinib once a day for 6-8 consecutive weeks of treatment，and receive ctDNA testing and radiographically imaging assessment again. According to test results, there are two types:

1. EGFR mutation is positive, subjects subsequent treament is up to the investigator (continue to receive 110 mg of Almonertinib once a day or combination therapy regimen), follow up every 6 weeks.
2. EGFR mutation is negative and achieve stable radiographically deep response after 6-8 weeks treatment with Almonertinib, subjects will stop Almonertinib treatment，and receive sequential Envafolimab immunotherapy (ctDNA dynamic monitoring guided treatment，every 6 weeks test ctDNA once, if it is negative, subjects continue to receive Envafolimab immunotherapy until ctDNA EGFR turns positive; if ctDNA EGFR is positive, subjects stop Envafolimab immunotherapy and receive Almonertinib 110 mg once a day again until ctDNA EGFR turns negative).

The treatment will continue until disease progression assessed by the investigator according to RECIST 1.1 criteria, or withdrawal or termination criteria are reached.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old (including 18 years old) .
* The Eastern Cooperative Oncology Group (ECOG) physical status score is 0 to 1, and it has not deteriorated in the previous 2 weeks, and the minimum expected survival is 12 weeks.
* Unresectable advanced or metastatic non-squamous cell non-small cell lung cancer.
* Blood samples were confirmed to contain EGFR-sensitive mutations by ctDNA testing(including exon 19 deletion or L858R, both alone or coexist with other EGFR mutations.Patients with EGFR20 exon insertion mutations could not be enrolled).
* No systematic antitumor treatment before enrollment.
* PD-L1 expression is positive, defined as TPS (tumor proportion score) ≥10%.
* The patient has at least one tumor lesion that can be accurately measured at baseline, and the longest diameter at baseline is ≥10 mm (if it is a lymph node, the short diameter is required to be ≥15 mm). The selected measurement method is suitable for accurate repeat measurement, which can be computed tomography (CT) or magnetic resonance scan (MRI). If there is only one measurable lesion, it can be accepted as the target lesion, and a baseline assessment of the tumor lesion should be performed at least 14 days after the diagnostic biopsy.
* Women of childbearing age should take appropriate contraceptive measures from screening to 3 months after stopping the study treatment and should not breastfeed. Before starting the administration, the pregnancy test is negative, or meeting one of the following criteria proves that there is no risk of pregnancy:

  1. Postmenopausal is defined as age greater than 50 years，and amenorrhea for at least 12 months after stopping all exogenous hormone replacement therapy.
  2. For women younger than 50 years old, if the amenorrhea is 12 months or more after stopping all exogenous hormone treatments, and the luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels are within the laboratory postmenopausal reference value range, also It can be considered postmenopausal.
  3. Have received irreversible sterilization, including hysterectomy, bilateral ovariectomy or bilateral fallopian tube resection, except for bilateral fallopian tube ligation.
* Male subjects should use barrier contraception (ie, condoms) from screening to 3 months after the study treatment is stopped.
* The subjects themselves participated voluntarily and signed a written informed consent form.

Exclusion Criteria:

Subjects who meet any of the following criteria cannot be included in this study:

* Have received any of the following treatments:

  1. Previously received antitumor treatment for lung cancer in the past;
  2. Previously received Chinese patent medicine with anti-tumor effect. If Chinese patent medicine with anti-tumor effect has been received for no more than 7 days, and the medicine has been stopped for 2 weeks or more before the drug treatment of this study, it can be included in the group.
* Patients who had received open surgery on other parts except lungs within 14 days before using the study drug ≤ 14 days.
* Refractory nausea, vomiting or chronic gastrointestinal diseases, inability to swallow the study drug or having undergone extensive intestinal resection may affect the full absorption of Almonertinib.
* Patients with other malignant tumors in recent 5 years (excluding completely resected basal cell carcinoma, bladder cancer in situ and cervical carcinoma in situ).
* Have a history of interstitial lung disease, a history of drug-induced interstitial lung disease, a history of interstitial pneumonia requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
* As judged by the investigator, there are any serious or poorly controlled systemic disease, such as poorly controlled hypertension, active bleeding or active infection (including active fungal, bacterial and / or viral infections requiring systemic treatment or full-body anti infective drugs used within one week before the first administration).
* At the beginning of the study treatment, there were unresponsive residual toxicity from previous treatment that was greater than CTCAE grade 3, except for hair loss.
* Meet any of the following cardiac examination results:

  1. The average value of QT interval (QTcF) corrected by Fridericia's formula obtained from 3 ECG examinations at rest> 470 msec;
  2. Resting ECG suggests that there are various clinically significant rhythms, conduction or ECG morphological abnormalities that are judged by the investigator (such as complete left bundle branch block, 3 degree atrioventricular block, 2 degree atrium Ventricular block and PR interval> 250 msec, etc.);
  3. There are any factors that increase the risk of QTc prolongation or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death or prolonged QT of immediate family members under 40 Any concomitant drugs in the interval;
  4. Left ventricular ejection fraction (LVEF) <50%.
* Insufficient bone marrow reserve or organ function, reaching any one of the following laboratory limits (no corrective treatment within 1 week before laboratory examination of blood draw):

  1. Absolute neutrophil count <1.5×109 / L; Platelet count <100×109 / L; Hemoglobin <90 g/L (<9 g/dL);
  2. Liver function: alanine aminotransferase > 3 times the upper limit of normal (ULN); Aspartate aminotransferase > 3uln; Total bilirubin > 1.5uln; Serum albumin (ALB) < 28 g / L.
  3. Renal function: creatinine > 1.5 ULN or creatinine clearance < 50ml / min (calculated by Cockcroft Gault formula). Only when creatinine ≥ 1.5 ULN, it is necessary to confirm creatinine clearance.
* Female subjects who are pregnant, lactating, or planning to become pregnant during the study period.
* Have a history of hypersensitivity to any active or inactive ingredients of almonertinib or to drugs with similar chemical structure to almonertinib or the same class of almonertinib.
* Any serious or uncontrolled eye disease (especially severe dry eye syndrome, dry keratoconjunctivitis, severe exposure keratitis or other diseases that may increase epithelial damage) may increase the safety of the patient by the doctor's judgment Sexual risk; or those with eye abnormalities that require surgery or are expected to require surgical treatment during the study period.
* Use / eat drugs or foods that are known to have strong CYP3A4 inhibition effect within 2 weeks (including but not limited to azanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nefenavir, ritonavir, saquinavir, telithromycin, acephaeomycin, voriconazole and grapefruit or grapefruit juice).
* Use drugs known to have strong CYP3A4 inducing effect (including but not limited to carbamazepine, phenobarbital, phenytoin, rifampin, rifampicin and Hypericum perforatum) within 2 weeks.
* Use drugs (including but not limited to dihydroergotamine, ergotamine, pimozide, astemizole, cisapride and terfenadine) as CYP3A4 substrates (with narrow therapeutic index) within 2 weeks.
* Have used strong P-gp inhibitors within 2 weeks (including but not limited to verapamil, cyclosporine A and dexverapamil)
* Patients with previous autoimmune diseases or undergoing immunomodulatory treatment.
* Subjects who may have poor compliance with the study procedures and requirements at the judgment of the investigator, such as those who have a clear history of neurological or mental disorders (including epilepsy or dementia) in the past, and those who currently suffer from mental disorders.
* Patients who need long-term systemic corticosteroids. Patients with COPD and asthma requiring intermittent use of bronchodilators, inhaled corticosteroids, or local injection of corticosteroids can be enrolled.
* Symptomatic central nervous system metastasis. Patients with asymptomatic brain metastases or brain metastases whose symptoms are stable after treatment can participate in this study as long as they meet all the following criteria: there are measurable lesions outside the central nervous system; No midbrain, pons, cerebellum, meninges, medulla oblongata or spinal cord metastasis; Maintain clinical stability for at least 2 weeks; Hormone therapy was stopped 3 days before the first dose of study drug.
* Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1 / 2 antibody positive).
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected is greater than the upper limit of the normal value of the laboratory of the research center); Note: hepatitis B subjects meeting the following criteria can also be included in the group:

  1. HBV viral load before the first administration was < 1000 copies / ml (200 IU / ml), and the subject should receive anti HBV treatment during the whole study chemotherapy drug treatment period to avoid virus reactivation;
  2. For subjects with anti HBC (+), HBsAg (-), anti HBS (-) and HBV viral load (-), preventive anti HBV treatment is not required, but viral reactivation needs to be closely monitored..
* Active HCV infected subjects (HCV antibody is positive and HCV-RNA level is higher than the lower limit of detection).
* Have received live vaccine within 30 days before the first administration (cycle 1, day 1); Note: it is allowed to receive inactivated virus vaccine for injection against seasonal influenza within 30 days before the first administration; subjects have received live attenuated influenza vaccine for intranasal administration is not allowed.
* Investigator judges that there are any patients with conditions that endanger the safety of the patient or interfere with the evaluation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months.
  The progression-free survival is defined as the time from date of baseline until the the date of first documented progression or date of death from any cause, whichever came first.
TRP | 24 months.
  Time to retest positive is defined as the time from date of sequential Envafolimab treatment until blood sample ctDNA detected for EGFR mutation recurrence or disease progression assessed by radiological imaging，assessed up to 24 months.

SECONDARY OUTCOMES:
ORR | From baseline, then every 6 weeks, until disease progression or discontinuation from study. ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression assessed up to 24 months.
  ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression, assessed up to 24 months.
DCR | 24 months.
  The disease control rate is defined as the proportion of patients with a best overall response of CR, PR, or SD.
OS | 24 months after the last subject participating in.
  OS is defined as the time from the starting date of study drug to the date of death，due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Qian Shu, Principal Investigator — Jiangsu Provincial People's Hospital; Wen Gao, Principal Investigator — Jiangsu Provincial People's Hospital; Pei Ma, Principal Investigator — Jiangsu Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No